CLINICAL TRIAL: NCT00529867
Title: A Randomized Open-Label Trial of the Efficacy of Artemether-Lumefantrine Suspension Compared With Artemether-Lumefantrine Tablets for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Children Less Than Five Years in Western Kenya
Brief Title: Randomised Efficacy Study of Two Artemether-Lumefantrine Oral Formulations for the Treatment of Uncomplicated P. Falciparum Malaria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dafra Pharma (Industry)
Collaborators: Kenya Medical Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSC protocol No. 1210
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Last update posted 2008-01-18 (Estimated); Status verified 2008-01

CONDITIONS: Malaria, Falciparum
Keywords: Artemether/Lumefantrine suspension; P. falciparum malaria; children; uncomplicated Plasmodium falciparum malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether; Lumefantrine; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Artemether/lumefantrine tablets
- B (Active Comparator)
  Interventions: Drug: Artemether/Lumefantrine suspension

INTERVENTIONS:
Drug: Artemether/lumefantrine tablets — Artemether/lumefantrine tablets containing 20mg artemether and 120mg lumefantrine
  Dosage: 5 - 14.9 kg: 1 tablet and 15 - 24.9 kg: 2 tablets
  Administered at 0, 8, 24, 36, 48, and 60 hours on days 0, 1, and 2
  Other Names: Coartem
  Arms: A
Drug: Artemether/Lumefantrine suspension — Artemether/lumefantrine suspension containing 15mg artemether and 90mg lumefantrine per 5ml suspension
  Dosage: 5.0 - 7.4 kg = 7 ml, 7.5 - 9.9 kg = 10 ml, 10 - 12.4 kg = 14 ml, 12.5 - 14.9 kg = 17 ml, 15 - 17.4 kg = 20 ml, 17.5 - 19.9 kg = 24 ml, 20 - 22.4 kg = 27 ml and 22.5 - 24.9 kg = 30 ml
  Administered once daily at 0, 24, and 48 hours on days 0, 1 and 2
  Other Names: Co-Artesiane suspension
  Arms: B

SUMMARY:
The purpose of this study is to compare the safety and efficacy in children aged 6 - 59 months with uncomplicated malaria, treated with either conventional artemether/lumefantrine tablets(Coartem®) or artemether/ lumefantrine suspension (Co-artesiane®) in Western Kenya

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 6 and 59 months
* Minimum body weight of 5kg
* Presence of fever (Temp >/= 37.5°C) or a history of fever in the last 24 hours
* Presence of asexual P. falciparum monoinfection
* Initial parasite density of between 2,000 and 200,000 asexual parasites/µl of blood
* Not suffering from severe and complicated forms of malaria
* Able to take drugs under study by the oral route
* Parent or guardian gives informed written consent to participate in study

Exclusion Criteria:

* Severe and/or complicated malaria (WHO, 2000 classification), including severe anaemia (Hb =/<5 g/dl), two or more seizures in last 24 hrs and hyper-parasitaemia (>200,000 µl)
* Patients treated with mefloquine, halofantrine within the 7 days before Day 0 or with quinine salts and artemisinin derivatives within 3 days before Day 0, or artemether-lumefantrine 30 days before Day 0
* Patients who require intensive care for malaria or another severe concomitant illness capable of interfering with the clinical evolution of malaria
* Patients with vomiting and/or diarrhoea
* Signs of severe malnutrition (defined as follows: children with weight/height ratio below 3 standard deviations or below 70% of the median of the WHO standardized reference values, or still with symmetrical oedema affecting both feet)
* Presence of general danger signs in children below 5 years or other signs of serious and complex Plasmodium falciparum, as stated in the present WHO definitions
* Patients with known history of heart disease or arrhythmia
* History of allergy to artemether/lumefantrine or quinine

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 267 (Actual)
Dates: Start 2007-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To compare PCR corrected cure-rates on day 14 and 28 | 1 year

SECONDARY OUTCOMES:
To determine and compare Adequate Clinical and Parasitological Response (ACPR) at days 14 and 28 | 28 days
To determine and compare proportion of children with gametocytes on days 0, 7, 14, and 28 | 28 days
Monitor any possible adverse reactions following use of both drugs | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Juma, Dr., Principal Investigator — Kenya Medical Research Institute
Locations (1):
- Chulaimbo Health Centre, Kisumu, Nyanza, Kenya

REFERENCES:
- [Derived] Belard S, Ramharter M, Kurth F. Paediatric formulations of artemisinin-based combination therapies for treating uncomplicated malaria in children. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD009568. doi: 10.1002/14651858.CD009568.pub2. PMID 33289099
- [Derived] Juma EA, Obonyo CO, Akhwale WS, Ogutu BR. A randomized, open-label, comparative efficacy trial of artemether-lumefantrine suspension versus artemether-lumefantrine tablets for treatment of uncomplicated Plasmodium falciparum malaria in children in western Kenya. Malar J. 2008 Dec 22;7:262. doi: 10.1186/1475-2875-7-262. PMID 19102746